CLINICAL TRIAL: NCT02275923
Title: Reveal LINQ™ Evaluation of Fluid
Acronym: REEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated as sufficient data was collected to determine if impedance measurements with the LINQ™ device could track body fluid changes.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REEF
Record Dates: First submitted 2014-10-17; First posted 2014-10-27 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (Experimental): 'Reveal LINQ™ Insertable Cardiac Monitor' will be used to measure changes in subject subcutaneous impedance and compare with the fluid status assessed by the volume removed from the hemodialysis subject during dialysis sessions.
  Interventions: Device: Reveal LINQ™ Insertable Cardiac Monitor

INTERVENTIONS:
Device: Reveal LINQ™ Insertable Cardiac Monitor — Insertable cardiac monitor

SUMMARY:
The purpose of this study is to investigate the use of subcutaneous impedance measured with an implanted Medtronic Reveal LINQ™ insertable cardiac monitor for use as a fluid status monitor in hemodialysis patients. The study will measure the changes in subject subcutaneous impedance and compare with the fluid status assessed by the volume removed from the hemodialysis subject during dialysis sessions. Subcutaneous impedance trends will also be evaluated between dialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who currently undergo in-clinic hemodialysis treatment prescribed 2 or 3 times per week
* Patients willing to be implanted with the Reveal LINQ™ device
* Patients greater than 21 years of age
* Patients willing and able to comply with the study procedures including giving informed consent

Exclusion Criteria:

* Patient has an active implanted cardiac medical device (e.g. IPG, ICD, CRT, etc)
* Patients who currently undergo home dialysis treatment
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager.
* Patient with a recent infection defined as 1) bacteremia within 60 days OR 2) (nonbacteremic) infection within 14 days
* Patient not suitable for Reveal LINQ™ implantation (e.g., severe cachexia, dermatologic conditions of the skin, or major medical or social conditions expected to reduce survival to < 6 months), in the opinion of the investigator

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (19.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  Australia | 7

OUTCOME MEASURES:

1. Primary Outcome: Average Fluid Volume Removed
Description: The average fluid volume removal during the dialysis session over all patients.
Time Frame: 24 Days
Population: Enrolled patients implanted with a LINQ device that had at least one dialysis session between 7 and 30 days post-implant. Formal statistical analysis was not performed because the likelihood from the pre-specified model did not converge due to small sample size. Average fluid loss is summarized instead.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Diagnostic
Number analyzed (Participants) | 6
mL | 2948 (683)

2. Primary Outcome: Change in Subcutaneous Impedance
Description: The change in impedance from the beginning to the end of a dialysis session, averaged over all patients and dialysis sessions
Time Frame: 24 days
Population: Patients implanted with a LINQ having at least one dialysis session between 7 and 30 days post-implant
Measure: Mean (Standard Deviation); unit: ohm
Arm/Group | Diagnostic
Number analyzed (Participants) | 6
ohm | 207 (97)

ADVERSE EVENTS:
Time Frame: Subjects were followed on average of 4.7 months with a range of 3 to 6 months.
Arm/Group | Diagnostic
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (N=7)
Conjunctivitis (Eye disorders) | 1 (1) — Patient presented to the Alfred Hospital with headache, fever and photophobia. Following admission and assessment he was diagnosed with conjunctivitis and discharged on the 28th July.
Arteriovenous fistula (Renal and urinary disorders) | 1 (1) — Post dialysis on the 20.01.15, a thrombosed AVF was diagnosed post ultrasound and was admitted to the Alfred Hospital for a planned fistulagram and plasty. He then required an extra dialysis session.
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) — Patient presented to Emergency with worsening abdominal pain. A abdominal CT scan showed ischemic bowel and an evolving small bowel obstruction. The subject underwent a laparotomy and small bowel resection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (N=7)
Application site anaesthesia (Surgical and medical procedures) | 1 (1) — Pt has complained of mild numbness and very occasional discomfort at the implant site since 11.04.15. R/w by Dr Scott Wilson and nil signs of infection or cause for concern. Patient happy to continue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No